CLINICAL TRIAL: NCT04302545
Title: Cystoinflation to Prevent Bladder Injury in Obstetrics and Gynaecology Surgery Part 1-Cystoinflation in Repeat C-section Part 2- Cystoinflation in Abdominal Hysterectomy Part3- Cystoinflation in Placenta Accreta Spectrum Management
Brief Title: Cystoinflation to Prevent Bladder Injury in Obstetrics and Gynaecology Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shazia Saaqib (Other)
Collaborators: King Edward Medical University (Other); Institute of Public Health, Pakistan (Other)
Responsible Party: Sponsor-Investigator, Shazia Saaqib, Assistant Professor Gynecology and Obstetrics, King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ERB#216/RC/KEMU; NCT#04302545 (Registry Identifier: Clinical trials.gov)
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Bladder Injury; Complications; Cesarean Section; Adhesions Pelvic

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned into cystoinflation group and control group after parallel assignment. In the cystoinflation group, the intervention will be retro-fill of the bladder with 300cc saline and clamping the drainage port of the catheter till the completion of adhesiolysis. In contrast, the urinary catheter of control group patients will be put on free drainage.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcome assessors are kept blind by just entering the random number assigned to the subject on the papers and notes are written without details of adhesiolysis. The completed outcome performas are sent to the assessors with the only random number entered and without the assigned group. The random number file is opened only after receiving results from the statistician. The care providers in theatre and principle surgeon cannot be blinded in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystoinflation group (Experimental): Bladder will be recognized by observing its gradual distension during bladder retro-fill with 300cc saline to perform adhesiolysis.
  Interventions: Procedure: Cystoinflation
- Control group (No Intervention): Pelvic adhesiolysis will be performed without bladder retrofill.

INTERVENTIONS:
Procedure: Cystoinflation — Bladder retrofill with 300cc saline to distend the bladder to recognize bladder outline
  Other Names: Bladder retrofill
  Arms: Cystoinflation group

SUMMARY:
Part1:The healthy pregnant women with previous operative deliveries admitted for elective C-section will be counselled and conditioned informed consent will be taken to be included in either study group if dense pelvic adhesions will be found during their operation. Adhesiolysis will be performed using bladder retro-fill with 300cc saline in the cystoinflation group, and without retro-fill in control.Both groups will be observed for bladder injury rate,bloodloss,operativetime,urinary tract infection,micturition problems and fistula formation.

Part2&3:Summary of Part 2 and 3 will be provided after publication

DETAILED DESCRIPTION:
Part1:Investigators will conduct this study to find the effectiveness of cystoinflation to prevent bladder injury in women with adhesions of previous C-sections. This prospective analytic longitudinal study will be conducted in Lady Willingdon Hospital, a tertiary care teaching hospital affiliated with King Edward Medical University Pakistan, from August 2017 to July 2019, after approval by the institutional review board of King Edward Medical University, Pakistan. The subjects will be randomly allocated to cystoinflation and control groups. The healthy pregnant women with previous operative deliveries admitted for elective C-section will be counselled and conditioned informed consent will be taken to be included in either study group if dense pelvic adhesions will be found during their operation. Adhesiolysis will be performed using bladder retro-fill with 300cc saline in the cystoinflation group, and without retro-fill in control. We will assess primary outcome by observing bladder injury rate, blood loss and operative time. The secondary outcome will be assessed by Urinary tract infection, micturition problems and fistula formation during 3month follow up period. The cystoinflation will be considered effective if the proportion of bladder injury in the study group will be less than 50% of the control group.

Part2&3:Details of part2&3 will be provided after publication

ELIGIBILITY:
Part1:Inclusion Criteria:

* • Healthy pregnant women of any age

  * Two or more previous C-sections
  * Gestational age between 38-40 weeks (confirmed by dating scan)
  * Dense Adhesions of Tulandi scores four or more.
  * women who give informed consent to participate in the study

Exclusion Criteria

:• Patients with medical disorders

* Bladder injury before group assignment
* Placenta previa
* Subjects experiencing micturition problems (dysuria, frequency, urgency, urinary retention, incontinence) before the study.

Eligibility criteria of part 2&3 will be provided after publication -

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — part1:Pregnant women Part2:Assigned to abdominal hysterectomy Part3:pregnant women with placenta accreta spectrum
Enrollment: 564 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Munazza Naheed, MBBS, Study Director — King Edward Medical University; Tayyaba Saeed, MBBS, Study Director — King Edward Medical University; Mohammad Khalid, MBBS, MHM, Study Director — Institute of Public Health, Pakistan
Locations (1):
- Lady Willingdon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No: There is no plan to make individual participant data available. The data will be made available to individual researchers on request after publication.

REFERENCES:
- [Result] O'Hanlan KA. Cystosufflation to prevent bladder injury. J Minim Invasive Gynecol. 2009 Mar-Apr;16(2):195-7. doi: 10.1016/j.jmig.2008.11.011. Epub 2009 Jan 9. PMID 19138575
- [Result] Pandey D, Mehta S, Grover A, Goel N. Indwelling Catheterization in Caesarean Section: Time To Retire It! J Clin Diagn Res. 2015 Sep;9(9):QC01-4. doi: 10.7860/JCDR/2015/13495.6415. Epub 2015 Sep 1. PMID 26500959
- [Result] Abdel-Aleem H, Aboelnasr MF, Jayousi TM, Habib FA. Indwelling bladder catheterisation as part of intraoperative and postoperative care for caesarean section. Cochrane Database Syst Rev. 2014 Apr 11;2014(4):CD010322. doi: 10.1002/14651858.CD010322.pub2. PMID 24729285
- [Result] Joelsson-Alm E, Nyman CR, Svensen C, Ulfvarson J. Micturition problems after bladder distension during hospitalization in Sweden: "I'm not ill, just damaged for the rest of my life". Nurs Res. 2014 Nov-Dec;63(6):418-25. doi: 10.1097/NNR.0000000000000057. PMID 25350541
- [Derived] Saaqib S, Naheed M, Iqbal A, Rehman RMAU, Khalid M. Evaluating a novel approach to placenta accreta spectrum management: the modified Triple-P technique with cystoinflation (a randomized controlled trial). Sci Rep. 2025 Jul 16;15(1):25870. doi: 10.1038/s41598-025-07582-6. PMID 40670452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in King Edward Medical University affiliated hospital/Lady Willingdon Hospital for a period of two years starting from August 1,2017 to July31,2019 including a 3month follow up period.
Pre-assignment Details: Subjects admitted with full term pregnancy and previous 2 C-sections n=734 The study subjects were selected in two step assessment(a)preoperative (during operation).
  preoperatively Excluded n=346 due to medical disorders, placenta previa, bladder injury before group assignment, micturition problems before operation Declined to participate=5 During operation Excluded=174 as criteria of dense adhesions of bladder was not met with.
Groups:
- Distension Arm: Subjects with no bladder injury
- Bladder Injury Arm: Subjects with bladder injury
Period: Overall Study
Arm/Group | Distension Arm | Bladder Injury Arm
Started | 107 | 107
Completed | 104 | 103
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: This study included Pakistani women eighteen years and above, coming to Lady Willingdon hospital for elective caesarean section due to the previous two or more C-sections, with no major medical disorder and found to have dense bladder adhesions on opening the abdomen; recognition of bladder was difficult due to overlying adhesions
Groups:
- Cystoinflation Group: Cystoinflation: Bladder will be retro-filled with 300cc saline to distend the bladder to recognize bladder outline in cystoinflation group whenever dense adhesions will be encountered which obscure the bladder either before or after opening the peritoneal cavity. Bladder outline will be recognized by observing its gradual distension during bladder retro-fill .The outcome of cystoinflation group will be divided into distension arm(no bladder injury arm) and bladder injury arm.
- Control Group: In control group,Pelvic adhesiolysis will be performed with bladder put on free drainage by urinary catheter.The outcome of control arm will be divided into distension arm(no bladder injury arm) and bladder injury arm.
- Total: Total of all reporting groups
Arm/Group | Cystoinflation Group | Control Group | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 107 | 214
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.19 (2.3) | 31.73 (2.4) | 31.96 (2.388)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 107 | 107 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Pakistan | 107 | 107 | 207
Parity [Count of Participants; unit: Participants]
  para2 | 35 | 33 | 68
  para3 | 60 | 60 | 120
  para4 | 10 | 10 | 20
  para5 | 2 | 4 | 6
BMI kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 30.73 (1.89) | 30.54 (1.86) | 30.635 (1.876)
Socioecnomic status [Count of Participants; unit: Participants]
  low (per capita family income <Rupees3000/month) | 39 | 41 | 80
  medium (per capita family income<Rupees3000-5000/month | 55 | 54 | 109
  high (per capita family income Rupees 5,000/month | 13 | 12 | 25
Number of previous C-sections [Count of Participants; unit: Participants]
  previous2 | 46 | 43 | 89
  previous3 | 52 | 54 | 106
  previous4 | 6 | 7 | 13
  previous5 | 3 | 3 | 6
Score of adhesions [Count of Participants; unit: Participants] — Dense adhesions were classified according to Tulandi score of adhesions. Adhesions less than 3cm scored 4. Adhesions between3-6cm scored as 8. Adhesion of .6cm scored as 16.
  Participants
    4 | 53 | 56 | 109
    8 | 38 | 36 | 74
    16 | 16 | 15 | 31
Preoperative postmicturition bladder volume [Median (Full Range); unit: ml] | 15 [10 to 30] | 20 [10 to 30] | 15 [10 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Bladder Injury Rate
Description: The bladder injury will be detected by direct visualization in the cesarean section before delivery of the baby during adhesiolysis of dense adhesions of the lower uterine segment, which cover and obscure the bladder. The bladder injury outcome will be measured as the number(percentage) of subjects with injury.
Time Frame: From the confirmation of adhesions to adhesiolysis and separation of bladder flap from uterus, before delivery of the baby during cesarean section.This time frame can range between 10-20 minutes.
Measure: Count of Participants; unit: Participants
Groups:
- Cystoinflation Group: Cystoinflation: Bladder retrofill with 300cc saline to distend the bladder to recognize bladder outline.
  Outcome will be studied as bladder injury arm and Distension arm
- Control Group: Pelvic adhesiolysis will be performed without bladder retrofill.Outcome will be studied as bladder injury arm and Distension arm.
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
Participants | 3 | 22
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Null Hypothesis: During the cesarean section of women with adhesions of the previous cesarean section that obscure the bladder, the bladder injury rate is not significantly decreased in cystoinflation group compared to the control. In this study, the bladder injury rate was seven times lesser in cystoinflation group compared to the control, thereby strongly supporting our hypothesis. The power of the study for bladder injury was 0.988, calculated with statistical software G'Power version 3.1; Test type: Other — Other Primary outcomes were the extent of injury, operative time, blood loss and proportion of subjects receiving a blood transfusion. Postoperatively, subjects were assessed for secondary outcomes of UTI, micturition problems, and fistula formation during the hospital stay and for the next 3 months. Postoperative micturition problems were feeling of incomplete evacuation, frequency, urgency, urethral and extra-urethral incontinence; p < .0001, Regression, Linear — The threshold for statistical significance was <.05; Odds Ratio (OR) = -.178, 95% CI 2-sided [-.261 to -.094]

2. Primary Outcome: Blood Loss
Description: Amount of blood loss during C-section will be increase in weight of sponges used during operation, taking 1gram equal to 1cc.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
ml | 585.32 (152.52) | 797.10 (385.09)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Odds Ratio (OR) = -211.776, 95% CI 2-sided [-290.70 to -132.84]

3. Primary Outcome: Operative Time
Description: Time from incision till closure of skin
Time Frame: During Caesarean section
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Cystoinflation Group: Bladder will be recognized by observing its gradual distension during bladder retro-fill with 300cc.
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
minutes | 45 (8.66) | 45 (16.99)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Null Hypothsis:Cystoinflation is ineffective to prevent bladder injury in adhesions of previous C-section.The cystoinflation was to be cosidered ineffective if proportion of bladder injury in study group was less than %0% of the control.The power of the study for bladder injury prevention was.988,calculated with statistical software G'Power version3.1; Test type: Other; p = 1, Regression, Linear; Odds Ratio (OR) = 0.000, 95% CI 2-sided [-3.634 to 3.634]

4. Secondary Outcome: White Blood Cells Count Per High Power Feild
Description: The normal white cell count ranges between 4000-11000 per microlitre. The raised count is an indication of postoperative infection.
Time Frame: 3rd postoperative day
Population: This analysis will be carried out in postoperative subjects of both groups.
Measure: Mean (Standard Deviation); unit: count/hpf
Groups:
- Cystinflation Group: Subjects in which adhesiolysis is performed after distending bladder with300cc saline.
- Control Group: Subjects in which adhesiolysis is performed with urinary catheter put on free drainage.
Arm/Group | Cystinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
count/hpf | 6.26 (1.003) | 7.36 (3.063)
Statistical Analysis 1: Comparison: Cystinflation Group vs Control Group; Test type: Other; p = .001, Regression, Linear; Odds Ratio (OR) = -1.093, 95% CI 2-sided [-1.708 to -.479]

5. Secondary Outcome: Urine Culture Report for Micro-organisms
Description: The outcome measure was the number(percentage) of subjects in which urine culture reports showed the growth of micro-organisms in the urine of the subjects sent for test on the second postoperative day.
Time Frame: 2nd postoperative day
Population: The population included all cases of both cystinflation group and control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
Participants | 2 | 18
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Odds Ratio (OR) = -.15, 95% CI 2-sided [-0.226 to -0.073]

6. Secondary Outcome: Fever
Description: Number of patients who presented with fever during hospital stay
Time Frame: upto 3months
Measure: Count of Participants; unit: Participants
Groups:
- Cystoinflation Group: Subjects in which adhesiolysis is performed after distending bladder with 300cc saline.
- Control Group: Subjects in which adhesiolysis is performed by putting urinary catheter on free drainage
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 107 | 107
Participants | 2 | 13
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p = 0.003, Regression, Linear; Odds Ratio (OR) = -.103, 95% CI 2-sided [-0.171 to -0.035]

7. Secondary Outcome: Postmicturition Bladder Volume After C-section
Description: Volume of urine retained in bladder after evacuation. Bladder distension will be diagnosed if volume retained in the bladder will be greater than 50cc measured on 4th postoperative day
Time Frame: upto 3months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
ml | 15.56 (4.968) | 14.91 (4.952)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p = .336, Regression, Linear; Odds Ratio (OR) = 0.654, 95% CI 2-sided [-0.682 to 1.991]

8. Secondary Outcome: Composite Micturition Problems During Hospital Stay
Description: The micturition problems during the hospital stay investigated in this study were dysuria, feeling of incomplete evacuation, frequency, urgency, urethral and extra-urethral incontinence), Dysuria was expressed by the subject as painful micturition using an 11point visual analogue Scale from zero to ten and converted into severity scores from 0-3.
  Score 0 or no point= 0 point on scale Score1 or mild pain=1-3point Score2 or Moderate Pain=4-6points; Score 3 or Severe Pain=.7-10 Other micturition problems (feeling of incomplete evacuation, frequency, urgency, urethral and extra-urethral incontinence) were measured subjectively on a 4point Likert scale questionnaire according to severity ranging from 0-3 (0-never, 1-rarely, 2-sometimes, and 3-often). The micturition problems of each subject were summed up as composite variables and both groups were compared for the mean value of the composite variable and standard deviation in spss20 statistical software.
Time Frame: Complaint recorded during hospital stay (range between 4-21 days)
Population: Subjects of both cystoinflation and control groups during the postoperative hospital stay.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
score | .077 (.633) | .47 (1.63)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p = .021, Regression, Linear; Odds Ratio (OR) = -0.393, 95% CI 2-sided [-0.725 to -0.06]

9. Secondary Outcome: Duration of Urinary Catheterization
Description: The time interval for which subject will be kept catheterized postoperatively.
Time Frame: upto 3months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
Days | 1.25 (1.626) | 3.14 (4.575)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p < 0.0001, Regression, Linear; Odds Ratio (OR) = -1.89, 95% CI 2-sided [-2.813 to -0.963]

10. Secondary Outcome: Duration of Hospital Stay
Description: The time interval in days from the date of operation till discharge from the hospital.
Time Frame: upto 3months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
Days | 4.18 (1.156) | 5.50 (3.506)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p < .0001, Regression, Linear; Odds Ratio (OR) = -1.318, 95% CI 2-sided [-2.021 to -0.614]

11. Secondary Outcome: Number of Subjects With Urinary Fistula Formation
Description: abnormal communication between genital tract nd urinary tract
Time Frame: upto 3months
Measure: Count of Participants; unit: Participants
Groups:
- Cystoinflation Group: The adhesiolysis will be carried out after retrograde bladder fill with 300cc saline.
- Control Group: The adhesiolysis will be carried out with urinary catheter put on free drainage.
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
Participants | 0 | 1

12. Secondary Outcome: Composite Micturition Problems After Discharge
Description: IT is composit Likert score(range from 0-3) of micturition problems recorded by patient after discharge from the hospital to the completion of 3months postoperative(follow up period).The lower value of the score is associated with good outcome while higher value shows a poor outcome.
Time Frame: upto 3months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Cystoinflation Group | Control Group
Number analyzed (Participants) | 104 | 103
score | .0047 (.034) | .0701 (.222)
Statistical Analysis 1: Comparison: Cystoinflation Group vs Control Group; Test type: Other; p = .003, Regression, Linear; Odds Ratio (OR) = -.065, 95% CI 2-sided [-.108 to -.023]

ADVERSE EVENTS:
Time Frame: Follow up was carried out over a period of 3months.
Description: Fortunately, there was no mortality as the population were young, healthy, adult women and all the women with medical disorders and surgical complications were excluded. The women with adhesions of previous C-section were at risk of bladder injury, excessive haemorrhage due to prolonged surgery..All the bladder injury cases were entered in the adverse event register of the study.
Arm/Group | Cystoinflation Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 3/107 | 22/107
Other Adverse Events (participants affected / at risk) | 0/107 | 1/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cystoinflation Group (N=107) | Control Group (N=107)
Bladder injury (Renal and urinary disorders) | 3 (3) | 22 (22) — abnormal communication between genital tract and urinary system
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cystoinflation Group (N=107) | Control Group (N=107)
vasicovaginal Fistula (Renal and urinary disorders) | 0 (0) | 1 (1) — injury to the urinary system during adhesiolysis of previous 2 or more C-sections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04302545/Prot_SAP_ICF_000.pdf